CLINICAL TRIAL: NCT03020823
Title: An Open-Label, Phase II Study to Evaluate the Efficacy and Safety of SCB01A in Subjects With Recurrent or Metastatic Squamous Cell Head and Neck Cancer Who Have Failed Platinum-Based Treatment
Brief Title: To Evaluate the Efficacy and Safety of SCB01A in Subjects With r/m Squamous Cell Head and Neck Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: withdrawal by sponsor
Sponsor: SynCore Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCB01A-22
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Results first posted 2023-06-02 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Head and Neck Neoplasms
Keywords: SCB01A; squamous cell carcinoma of head and neck
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — indole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SCB01A alone (Experimental): intra-subject dose escalation starting from 12 mg/m2, then to18 mg/m2, and finally to 24 mg/m2 if no DLT
  Interventions: Drug: SCB01A

INTERVENTIONS:
Drug: SCB01A — intra-subject dose escalation, 12, 18, 24 mg/m2, 24h-IV infusion (in the vein) on day 1 and 8 of each 21 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: 6-Methoxy-3-(3',4',5'-trimethoxybenzoyl) indole

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of i.v. infusion for 24-hour of SCB01A in subjects with squamous cell carcinoma of head and neck who have failed previous platinum based therapies.

DETAILED DESCRIPTION:
From pre-clinical pharmacology and phase I clinical study SCB01A has demonstrated promising anticancer action with a vascular disrupting activity that has the potential for treatment of various malignancies, particularly for patients with drug resistance. The drug has been studied in human subjects in a dose escalation phase I study and has shown to be safe for up to 2 cycles of 24 mg/m2 (each cycle consisting of one intravenous [i.v.] administration of SCB01A via a central line every 3 weeks). In the phase I study, partial response (PR) (shrinkage of tumor size to 50%) was observed in cycle 9 (3 mg/m2) of one subject with right buccal squamous cell carcinoma and 19/33 (58%) subjects had stable disease (SD) for more than 2 cycles.

Pre clinical study of SCB01A showed that the concentrations at which tubulin inhibition occurred were around 80 nM for 24-hour exposure or 200 nM for 6-hour exposure. However, pharmacokinetic (PK) results of phase I study showed that the average elimination half-life (t1/2) of a 3-hours i.v. infusion of SCB01A is approximately 2.5 hours and almost no SCB01A can be detected after 10 hours, indicating most subjects were treated in short API exposure time and may have been insufficient to achieve efficacy. Therefore, to extend the exposure duration above effective concentration in blood may increase the treatment efficacy.

The aim of this study is to evaluate the efficacy and safety of i.v. infusion for 24-hour of SCB01A in subjects with squamous cell carcinoma of head and neck who have failed previous platinum based therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥20 years;
2. Signed informed consent obtained prior to initiation of any study-specific procedures and treatment;
3. Histological or cytological confirmed squamous cell carcinoma of head and neck, excluding nasopharyngeal carcinoma;
4. Subjects with unresectable, unfeasible radiotherapy, recurrent or metastatic head and neck squamous cell carcinoma, after previous treatment with platinum agent;
5. Subjects must have at least one measurable tumor lesion as defined by RECIST version 1.1 as assessed by the investigator (local radiological image assessment) or clinically evaluable disease. Physical and neurological examinations, and radiographic studies have to be performed within 28 days of Cycle 1 Day 1;
6. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-1;
7. Life expectancy of 12 weeks or longer;
8. Concurrent local therapy is not allowed, but concurrent palliative radiation therapy to non-measurable sites of disease such as painful bone metastasis is permitted;
9. All eligible subjects of childbearing potential have to use effective contraception; that is, double barrier contraceptive methods;
10. Documented progressive disease within past 6 months;
11. Adequate bone marrow reserve, cardiac, renal and liver function:

    1. Absolute neutrophil count (ANC) > 1.5 x 109/L;
    2. White blood cell (WBC) > 3 x 109/L;
    3. Platelet count > 75 x 109/L;
    4. Hemoglobin > 9 g/dL ( > 5.6 mmol/l);
    5. Prothrombin time (PT)/international normalized ratio (INR) ≤1.5 x upper limit of normal (ULN);
    6. Creatinine clearance (Cockcroft & Gault formula) >50 mL/min;
    7. Alanine aminotransferase (ALT, SGPT) and aspartate aminotransferase (AST, SGOT) and Alkaline Phosphatase (ALP) < 3 x ULN; AST/ALT≦5 x ULN if liver metastasis;
    8. Serum albumin ≥ 3 g/dL;
    9. Total Bilirubin ≤ 1.5 x ULN;
    10. QTc <450 msec

Exclusion Criteria:

1. Known primary CNS malignancy or CNS involvement (except for brain metastases that have been treated and are stable and subject is off steroids);
2. Chemotherapy, radiation therapy, major surgery or investigational agents including immune or target therapies less than 4 weeks prior to study drug treatment;
3. History of malignancy other than head and neck cancer with the exception of early stage non-melanoma skin cancer or carcinoma in situ of cervix;
4. History of liver cirrhosis;
5. Active hepatitis B or hepatitis C infection;
6. Clinical significant pulmonary obstructive or clinical significant pulmonary restrictive diseases (grade >2);
7. Clinically significant cardiac disease (NYHA class > 2);
8. Other serious illness or medial conditions, such as active infection, unresolved bowel obstruction, or psychiatric disorders;
9. Known HIV positivity;
10. Pregnant or breast-feeding subjects, and men and women of child-bearing potential not using effective contraception while on study treatment;
11. Known hypersensitivity to any component of SCB01A or excipients including Solutol®, alcohol, and PEG300;
12. History of exposure to SCB01A or its analogues;
13. History of active or significant neurological disorder or psychiatric disorder that would prohibit the understanding and giving of informed consent, or would interfere with the clinical and radiological evaluation of central nervous system during the trial;
14. Peripheral neuropathy (≥ grade 2);
15. Any other reason the investigator deems the subject to be unsuitable for the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-04-30 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Her-Shyong Shiah, MD, Principal Investigator — Taipei Medical University Hospital
Locations (4):
- Taiwan (4):
  - National Cheng Kung University Hospital, Tainan
  - Suang Ho Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intra-subject Dose Escalation Regimen: All subjects enrolled in this study would be treated from the same starting dose 12 mg/m² (Dose 1) given on Days 1 and 8 in a 21-day cycle by 24 h i.v. infusion. If the subject experiences no dose-limiting toxicity (DLT) during the period, dose escalation of SCB01A to 18 mg/m² (Dose 2) occurred from cycle 2; and increased to 24 mg/m² (Dose 3) on cycle 3.
Period: Overall Study
Arm/Group | Intra-subject Dose Escalation Regimen
Started | 10
12 mg/m² Only | 3
12 & 18 mg/m² | 4
12, 18 & 24 mg/m² | 3
Completed | 0 (4 subjects discontinued from the study owing to disease progression based on clinical judgement, 4 subjects discontinued because of diagnosed PD based on RECIST, and 2 subjects discontinued because of intolerable adverse event(s) or failure to tolerate the study treatment.)
Not Completed | 10
Not completed — Physician Decision | 4
Not completed — Lack of Efficacy | 4
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | SCB01A Alone
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 10
Region of Enrollment [Number; unit: participants]
  Taiwan | 10
ECOG at Screening visit [Count of Participants; unit: Participants] — ECOG 0: Normal activity. Fully active, able to carry on all pre-disease performance without restriction.
  ECOG 1: Symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work).
  Participants
    0 | 4
    1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) During Treatment Phase
Description: Objective response rate (ORR) was defined as complete response (CR) + partial response (PR), according to RECIST v1.1 criteria.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to approximately 15 months (assessed continuously during treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | SCB01A Alone
Number analyzed (Participants) | 10
Participants | 0

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from the start of treatment up to the date of first progression based on RECIST v1.1 or the date of death, which ever comes first.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: From the start of treatment up to either first observation of progressive disease or occurrence of death, up to approximately 15 months (assessed continuously during treatment)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | SCB01A Alone
Number analyzed (Participants) | 10
days | 125 [28 to 251]

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the as the time from the start of treatment up to the time that the subject is still alive.
Time Frame: From the start of treatment up to death from any cause or last day known to be alive, up to approximately 15 months (assessed continuously during treatment)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | SCB01A Alone
Number analyzed (Participants) | 10
days | 292 [29 to 292]

4. Secondary Outcome: Best Overall Tumor Response
Description: Best overall tumor response is defined as an objective response or stable disease of treatment phase.
Time Frame: Up to approximately 15 months (assessed continuously during treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | SCB01A Alone
Number analyzed (Participants) | 10
Participants | 3

ADVERSE EVENTS:
Time Frame: Up to approximately 15 months (assessed continuously during treatment)
Groups:
- SCB01A 12 mg/m² Only; SCB01A 12 & 18 mg/m²; SCB01A 12, 18 & 24 mg/m²: All subjects enrolled in this study would be treated from the same starting dose 12 mg/m² (Dose 1) given on Days 1 and 8 in a 21-day cycle by 24 h i.v. infusion. If the subject experiences no dose-limiting toxicity (DLT) during the period, dose escalation of SCB01A to 18 mg/m² (Dose 2) occurred from cycle 2; and increased to 24 mg/m² (Dose 3) on cycle 3.
Arm/Group | SCB01A 12 mg/m² Only | SCB01A 12 & 18 mg/m² | SCB01A 12, 18 & 24 mg/m²
All-Cause Mortality (participants affected / at risk) | 2/3 | 2/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/4 | 0/3
Other Adverse Events (participants affected / at risk) | 2/3 | 4/4 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCB01A 12 mg/m² Only (N=3) | SCB01A 12 & 18 mg/m² (N=4) | SCB01A 12, 18 & 24 mg/m² (N=3)
somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCB01A 12 mg/m² Only (N=3) | SCB01A 12 & 18 mg/m² (N=4) | SCB01A 12, 18 & 24 mg/m² (N=3)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Edema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ear injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Ear neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (4):
  • Study Protocol (2016-12-19): https://cdn.clinicaltrials.gov/large-docs/23/NCT03020823/Prot_000.pdf
  • Statistical Analysis Plan: TableFigure (2018-12-14): https://cdn.clinicaltrials.gov/large-docs/23/NCT03020823/SAP_001.pdf
  • Statistical Analysis Plan: Listing (2018-12-14): https://cdn.clinicaltrials.gov/large-docs/23/NCT03020823/SAP_002.pdf
  • Statistical Analysis Plan: CSR_9.7_Statistical methods planned in the protocol (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/23/NCT03020823/SAP_003.pdf